CLINICAL TRIAL: NCT01412619
Title: CSINVOS: Non-invasive Measurement of Regional Intracerebral Tissue Oxygenation in Elective Cardiac Surgeries
Brief Title: Non-invasive Measurement of Regional Intracerebral Tissue Oxygenation in Elective Cardiac Surgeries
Acronym: CSINVOS
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: PI: PD Dr. med. Steffen Rex, Clinic for Anaesthesiology, Clinical Trial Center Aachen
Other Study IDs: CTC-A 11-131 CSINVOS
Record Dates: First submitted 2011-08-02; First posted 2011-08-09 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Neurological Outcome
Keywords: Neurological Outcome; Intraoperative intracerebral Oxygen level; Mean arterial blood pressure; Central venous blood pressure; Cardiac output; Serum Lactate; Venous oxygen saturation; Fluid balance

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cytokine IL-6 Cytokine IL-10 Procalcitonin (PCT) S-100-Protein
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients after cardiac surgical operations often exhibit neuropsychological complications. In particular, the post-operative delirium is associated with a significantly increased morbidity and mortality.

Intracerebral microembolization in addition to inadequate cerebral perfusion during surgery was verified as the main cause of this.

The aim of the study is to demonstrate a correlation between intraoperative low measured cerebral oxygen levels and a loss neurological outcome, especially the development of postoperative delirium, using non-invasive cerebral oximetry (RSO2).

DETAILED DESCRIPTION:
Before the operation, the parameters required for the collection of the EURO-scores are recorded, allowing an assessment of perioperative risk (age, gender, type of planned surgery, concomitant diseases).

After the patient arrives in the operating room the required electrodes to measure the intracerebral oxygenation are stuck bitemporal on the patient´s head. The measurement of oxygenation begins before induction of anaesthesia (while the patient is still awake) and will continue until 24 h postoperatively.

The measurement of cerebral oxygenation is not intended to serve as a replacement for the collection of routine peripheral oxygen saturation, but will be performed additionally.Therefore the anaesthesiological management depends primarily on the peripheral oxygen saturation and arterial blood gases according to our clinical routine.

If, however, intracerebral oxygenation shows an ominous decline, this change can be corrected by targeted measures very early (such as increasing the inspiratory oxygen concentration). At the specified test points following additional parameters are determined: Mean arterial blood pressure, central venous blood pressure, cardiac output, serum lactate, venous oxygen saturation, arterial blood gas analysis, fluid balance. These parameters are collected as part of a routine cardiac surgery. To measure these parameters no additional punctuation or blood draws are therefore necessary. To determine the cytokines IL-6 and IL-10, procalcitonin (PCT) and the S-100 protein, however, it is necessary to take 5ml blood to the respective measuring points from an already existing venous access.

In the ICU the collection of the above mentioned parameters occurs at admission, after 6h and 12h, and on the morning of the first postoperative day (and possibly on further ICU-treatment-days). Additionally, each 12 h after surgery, the SOFA and the CAM-ICU-Score are recorded.

An already before surgery performed CAM-ICU questionnaire serves as a direct comparison with the post-operative acquired CAM-ICU score. In case the patient is still be ventilated, the test cannot be performed and will be documented correspondingly.

The treatment, monitoring of vital signs including intermittent blood gas analysis and other diagnostic measures (clinical chemistry, radiology, etc.) corresponds to the standard surgical procedure for heart surgery of the University Hospital Aachen.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Elective cardiac surgery at heart-lung-machine

Exclusion Criteria:

* Pregnancy or lactation period
* Patients not capable of consenting
* Emergency surgery
* Patients under 18 years
* Known depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 100 adult patients (male and female), capable of consenting, undergoing elective cardiac surgery at heart-lung-machine
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
CAM-ICU (Confusion Assessment Method for the Intensive Care Unit) Questionnaire | Changes between 6 - 48 hours before surgery and 12 hours after surgery
  CAM-ICU Quesionnaire is used to assess the patient´s ability of postoperative orientation, to detect and treat changes between preoperative and postoperative questionnaires and therefore a potential postoperative delirium earliest possible.

SECONDARY OUTCOMES:
MIF (Macrophage Migration Inhibitory Factor) | Preoperative (2-30 minutes) after induction of anaesthesia, but (2-30 minutes) before starting surgery and postoperative immediately after admission to ICU, 4 hours after admission and every further morning in ICU in context of routine blood tests.
  MIF is used as inflammatory marker to ensure an uncomplicated postoperative period and to be able to react appropiately in case of values outsite expected range.
Cytokine IL-6 | Preoperative (2-30 minutes) after induction of anaesthesia, but (2-30 minutes) before starting surgery and postoperative immediately after admission to ICU, 4 hours after admission and every further morning in ICU in context of routine blood tests.
  Cytokine IL-6 is used as inflammatory marker to ensure an uncomplicated postoperative period and to be able to react appropiately in case of values outsite expected range.
Cytokine IL-10 | Preoperative (2-30 minutes) after induction of anaesthesia, but (2-30 minutes) before starting surgery and postoperative immediately after admission to ICU, 4 hours after admission and every further morning in ICU in context of routine blood tests.
  Cytokine IL-10 is used as inflammatory marker to ensure an uncomplicated postoperative period and to be able to react appropiately in case of values outsite expected range.
Procalcitonin (PCT) | Preoperative (2-30 minutes) after induction of anaesthesia, but (2-30 minutes) before starting surgery and postoperative immediately after admission to ICU, 4 hours after admission and every further morning in ICU in context of routine blood tests.
  PCT is used as inflammatory marker to ensure an uncomplicated postoperative period and to be able to react appropiately in case of values outsite expected range.
S-100 Protein | Preoperative (2-30 minutes) after induction of anaesthesia, but (2-30 minutes) before starting surgery and postoperative immediately after admission to ICU, 4 hours after admission and every further morning in ICU in context of routine blood tests.
  S-100 Protein is used as inflammatory marker to ensure an uncomplicated postoperative period and to be able to react appropiately in case of values outsite expected range.
SOFA-Score (Sequential Organ Failure Assessment score) | 12 hours after surgery
  The SOFA score is used to track a patient's status during the stay in the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Aachen, Aachen, Germany

REFERENCES:
- [Derived] Stoppe C, Fries M, Rossaint R, Grieb G, Coburn M, Simons D, Brucken D, Bernhagen J, Pallua N, Rex S. Blood levels of macrophage migration inhibitory factor after successful resuscitation from cardiac arrest. PLoS One. 2012;7(4):e33512. doi: 10.1371/journal.pone.0033512. Epub 2012 Apr 10. PMID 22506003